CLINICAL TRIAL: NCT01277094
Title: Multi-center, Double-blind, Randomized, Placebo-controlled Study of Selective 11 Beta-HSD1 Inhibition With RO5093151 for 12 Weeks to Investigate Efficacy, Safety and Pharmacokinetics of RO5093151 in Non-alcoholic Fatty Liver Disease and Its Metabolic Consequences.
Brief Title: A Study of RO5093151 in Patients With Non-Alcoholic Fatty Liver Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: BP25414
Record Dates: First submitted 2011-01-13; First posted 2011-01-14 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Fatty Liver, Non-alcoholic Fatty Liver Disease, NAFLD
MeSH Terms: conditions — Fatty Liver; Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: RO5093151
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Oral daily doses for 12 weeks
  Arms: 2
Drug: RO5093151 — Oral daily doses for 12 weeks
  Arms: 1

SUMMARY:
This multi-center, double-blind, randomized, placebo-controlled study will evaluate the change in liver fat content, pharmacokinetics and safety of RO5093151 in patients with non-alcoholic fatty liver disease. Patients will be randomized to receive either daily oral doses of RO5093151 or matching placebo. The anticipated time on study treatment is 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, 35-65 years of age
* Hepatic steatosis assessed by magnetic resonance spectroscopy (MRS) with liver fat >5.56% at screening
* Body mass index (BMI) >27 kg/m2 at screening
* Insulin resistance assessed by homeostatic model assessment-insulin resistance (HOMA-IR) > 2.5 at screening
* Agreement to maintain prior diet and exercise habits during the full course of study

Exclusion Criteria:

* History of diabetes mellitus based on World Health Organization (WHO) criteria
* Known polycystic ovary syndrome
* Other liver disease e.g. chronic viral hepatitis, alcoholic liver disease, hemachromatosis, cirrhosis
* Known autoimmune disease or chronic inflammatory disease
* Myocardial infarction or stroke within 6 months prior to screening
* Patients taking any anti-diabetic and/or weight-lowering medication currently or within the previous 3 months before screening

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2011-04; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Change of liver fat content measured by magnetic resonance spectroscopy (MRS) | Week 12

SECONDARY OUTCOMES:
Change in insulin resistance assessed by hyperinsulinemic euglycemic clamp | Week 12
Change in endogenous glucose production assessed by hyperinsulinemic euglycemic clamp | Week 12
Pharmacokinetic measures (max and min concentration, clearance, half-life, etc) | Week 12
Safety (incidence and nature of adverse events) | Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (4):
- Vienna, Austria
- Germany (3):
  - Düsseldorf
  - Nuthetal
  - Tübingen

REFERENCES:
- [Derived] Stefan N, Ramsauer M, Jordan P, Nowotny B, Kantartzis K, Machann J, Hwang JH, Nowotny P, Kahl S, Harreiter J, Hornemann S, Sanyal AJ, Stewart PM, Pfeiffer AF, Kautzky-Willer A, Roden M, Haring HU, Furst-Recktenwald S. Inhibition of 11beta-HSD1 with RO5093151 for non-alcoholic fatty liver disease: a multicentre, randomised, double-blind, placebo-controlled trial. Lancet Diabetes Endocrinol. 2014 May;2(5):406-16. doi: 10.1016/S2213-8587(13)70170-0. Epub 2014 Feb 17. PMID 24795254